CLINICAL TRIAL: NCT03025750
Title: Safety and Immunogenicity of Adjuvanted Reduced Dose Inactivated Polio Vaccine, IPV-Al SSI, in Comparison to Non-adjuvanted Full Dose IPV SSI, in Infants Vaccinated at 2, 4 and 6 Months of Age
Brief Title: Safety and Immunogenicity of Adjuvanted Reduced Dose Inactivated Polio Vaccine in 2, 4, 6 Months of Age
Acronym: VIPV-07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Larix A/S (Industry); Vaxtrials S.A. (Other); AJ Vaccines A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VIPV-07
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPV-Al SSI (Experimental): IPV-Al contains the reduced dose of IPV to be administered intramuscularly to the anterolateral of the right thigh. Each subject randomised to this group will receive a total of three primary injections - one at 2 months, 4 months and 6 months of age.
  Interventions: Biological: IPV-Al SSI
- IPV SSI (Active Comparator): IPV SSI contains the full dose of IPV to be administered intramuscularly to the anterolateral of the right thigh. Each subject randomised to this group will receive a total of three primary injections - one at 2 months, 4 months and 6 months of age.
  Interventions: Biological: IPV SSI

INTERVENTIONS:
Biological: IPV-Al SSI — Total of three primary injections of IPV-Al SSI, one at 2, 4 and 6 months of age
  Arms: IPV-Al SSI
Biological: IPV SSI — Total of three primary injections of IPV SSI, one at 2, 4 and 6 months of age
  Other Names: IPV Vaccine SSI
  Arms: IPV SSI

SUMMARY:
The trial is a phase III, non-inferiority, observer-blind, randomised, active controlled, multicentre clinical trial with 2 parallel groups: IPV-Al SSI (investigational vaccine) and IPV SSI (comparator vaccine). The vaccines will be administered at 2, 4 and 6 months of age.

DETAILED DESCRIPTION:
In addition to the trial vaccines (IPV-Al SSI or IPV SSI), the trial subjects will receive concomitant childhood vaccinations during the trial period. The trial vaccine (IPV-Al SSI or IPV SSI) is administered in the RIGHT thigh, whereas the other injectable childhood vaccines are administered in the opposite (LEFT) thigh.

At Visit 1 (inclusion, screening, blood sample, randomisation and 1st vaccination), written informed consent is obtained and the subject's eligibility is assessed according to the pre-specified in-/exclusion criteria. Information on medical history, demographics and concomitant medication are collected and a physical examination is performed and vital signs are measured. A prevaccination blood sample is taken for polio antibody determinations and the subject is randomly allocated into one of the two vaccination groups and vaccinated. A subset of 200 subjects are randomly chosen to have an extra blood sample taken at Visit 3. The subject is observed for immediate AEs 30 minutes after all vaccinations. An eDiary, thermometer and ruler are handed out to the parents for measurements of temperature and recording of injection site reactions and solicited systemic AEs. These activities are performed daily, starting on the day of the vaccination and the following 2 days and until resolved, and for recording of any other AEs as instructed by the trial staff. A contact to the parents via telephone will be made after the vaccination visit to remind the parents to fill in the eDiary and to check if they have any questions regarding how use the eDiary.

At Visit 2 (2nd vaccination), 2 months after Visit 1, the eDiary is collected and AEs and concomitant medications are recorded. Contraindications are reviewed, the 2nd vaccination is administered, immediate reactions are observed and the eDiary is returned to the partents for recordings of AEs and concomitant medications. A contact to the parents via telephone will be made after the vaccination visit to remind the parents to fill in the eDiary and to check if they have any questions regarding how use the eDiary.

At Visit 3 (3rd vaccination), 2 months after Visit 2, the eDiary is collected and AEs and concomitant medication are recorded. A blood sample from a subset of the subjects is taken for polio antibody determinations. Contraindications are reviewed, the 3rd vaccination is given, immediate reactions are observed and the eDiary is returned to the parents. A contact to the parents via telephone will be made after the vaccination visit to remind the parents to fill in the eDiary and to check if they have any questions regarding how use the eDiary.

At Visit 4 (blood sample and trial completion), 1 month after Visit 3, the eDiary is collected and AEs and concomitant medications are recorded and a blood sample for polio antibody determination is taken.

A safety follow-up telephone call will be conducted at 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants 2 months of age (54-75 days of age) on date of first vaccination
* Healthy assessed from medical history and physical examination
* Parent(s)/guardian(s) have been properly informed about the trial and signed informed consent form
* Parent(s)/guardian(s)granted access to the infant's trial related medical records
* Parent(s)/guardian(s)are likely to comply with trial procedures

Exclusion Criteria:

* Vaccinated with any polio vaccine other than the trial vaccines, prior to inclusion or planned during the trial
* OPV vaccination or known exposure to poliovirus (wild or vaccine-derived) in household (living together) within 3 months prior to inclusion or planned during the trial
* Low birth weight (< 2,500 g)
* Known or suspected immunodeficiency (e.g. leukaemia, lymphoma) or family history of congenital or hereditary immunodeficiency. HIV infection is not an exclusion criteria
* Severe uncontrolled chronic (e.g. neurologic, pulmonary, gastrointestinal, hepatic, renal or endocrine) disease
* Known or suspected allergy to vaccine constituents (e.g. hypersensitivity to formaldehyde, aluminium or 2-phenoxyethanol)
* Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections or blood sampling
* Treatment with a product which is likely to modify the immune response (e.g. systemic corticosteroids, blood products and immunoglobulins) prior to inclusion or planned during the trial period
* Participating in another clinical trial
* Not suitable for inclusion in the opinion of the investigator

Ages: 54 Days to 75 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Seroconversion for poliovirus type 1, 2 and 3 for IPV-Al compared to IPV SSI in infants | Change from baseline to one month after 3rd vaccination

SECONDARY OUTCOMES:
Adverse events following vaccinations (key secondary) | After primary injections at 2, 4 and 6 months of age
Subjects with seroprotection against poliovirus types 1, 2 and 3 | One months after 3rd vaccination
Subjects with poliovirus types 1, 2 and 3 post-vaccination titres >= 4-fold above estimated titre of maternal antibody | One months after 3rd vaccination
Geometric mean titres (GMTs) and median titers for poliovirus types 1, 2 and 3 | One months after 3rd vaccination
Reverse cumulative titre distribution curves for poliovirus types 1, 2 and 3 | From baseline and one months after 3rd vaccination

OTHER OUTCOMES:
Subject with seroconversion against poliovirus types 1, 2 and 3 | Two months after 2nd vaccination
Subjects with seroprotection against poliovirus types 1, 2 and 3 | Two months after 2nd vaccination
Subjects with poliovirus types 1, 2 and 3 post-vaccination titres ≥ 4-fold above estimated titre of maternal antibody | Two months after 2nd vaccination
Geometric mean titres (GMTs) and median titers for poliovirus types 1, 2 and 3 | Two months after 2nd vaccination
Reverse cumulative titre distribution curves for poliovirus types 1, 2 and 3 | From baseline and two months after 2nd vaccination
Sensitivity analysis: subjects with ≥ 4-fold increases in poliovirus types 1, 2 and 3 titres | From baseline and one months after 3rd vaccination
Sensitivity analysis: sub-groups of subjects with seroprotection (titre ≥ 8) and without seroprotection (titre < 8) at baseline | One months after 3rd vaccination
  * Subjects with seroconversion against poliovirus types 1, 2 and 3
  * Subjects with seroprotection (titre ≥ 8) against poliovirus types 1, 2 and 3
  * Subjects with poliovirus types 1, 2 and 3 post-vaccination titres ≥ 4-fold above the estimated titre of maternal antibody
  * Geometric mean titres (GMTs) and median titers for poliovirus types 1, 2 and 3
  * Reverse cumulative titre distribution curves for poliovirus types 1, 2 and 3 at baseline and one month after 3rd vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Kromann, Study Director — Statens Serum Institut
Locations (1):
- Cevaxin, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saez-Llorens X, Thierry-Carstensen B, Stoey LS, Sorensen C, Wachmann H, Bandyopadhyay AS, Nielsen PI, Kusk MV. Immunogenicity and safety of an adjuvanted inactivated polio vaccine, IPV-Al, following vaccination in children at 2, 4, 6 and at 15-18 months. Vaccine. 2020 May 6;38(21):3780-3789. doi: 10.1016/j.vaccine.2020.02.066. Epub 2020 Apr 6. PMID 32273184